CLINICAL TRIAL: NCT02695914
Title: Inflammatory Markers in Patient of FUO With Excess-heat Syndrome and the Influence of Compound Qingre Granule on the Inflammatory Markers
Brief Title: Influence of Compound Qingre Granule on the Inflammatory Markers in Patient of FUO With Excess-heat Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Miao Shi, postgraduate, Beijing Friendship Hospital
Other Study IDs: JJ2015-49
Record Dates: First submitted 2016-01-31; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Fever of Unknown Origin
Keywords: Inflammatory markers
MeSH Terms: conditions — Fever of Unknown Origin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Exsanguinating and saving the blood in the refrigerator of -4 ℃.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Conventional treatment methods will be given to cases in control group.
- Experiment group: On the base of control group, Compound Qingre Granule will be added to in experiment group.
  Interventions: Drug: Compound Qingre Granule

INTERVENTIONS:
Drug: Compound Qingre Granule — A kind of Chinese patent medicine, which is developed by Dr.Shuwen Zhang and Dr.Baoen Wang from Beijing Friendship Hospital.
  Other Names: Fufang Qingre Keli
  Groups: Experiment group

SUMMARY:
The purpose of this study is to observe inflammatory markers like TNF (tumor necrosis factor), IL-1 (interleukin-1), IL-6 (interleukin-6),TREM-1 (triggering receptor expressed on myeloid cells-1), etc, in patient of FUO with excess-heat syndrome and the influence of Compound Qingre Granule on the inflammatory markers.

DETAILED DESCRIPTION:
All the cases will be provided by the Infectious Diseases Department of Beijing Friendship Hospital.Each patient should sign informed consent. Assessing the accuracy, completeness, or representativeness of registry data by comparing the data to medical records. After collecting, sorting and entering the data, reducing the missing value, and then checking into the database.

The stochastic indicator method will be used to simple random sampling, to ensure the probabilities of each individuals be given Chinese medicine intervention are equal.Operations must be standard to reduce errors.

Quality assurance plan: Patient of fever within two weeks, or whose temperature is below 38.5 degree centigrade will be excluded. The registration form includes the following parts: Name, sex, age, address, phone number, admission time, primary diagnoses and levels of Inflammatory markers.

Data will be analyzed using the SPSS17.0 (Statistical Product and Service Solutions 17.0) statistical software. Difference of measurement data will be compared with analysis of variance,and difference of enumeration data will be compared with rank-sum test.P<0.05 has statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patient of fever of unknown origin (FUO).

Exclusion Criteria:

* Patient of fever within two weeks, or whose temperature is below 38.5 degree centigrade.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient of fever of unknown origin with excess-heat syndrome
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Inflammatory marker (TREM-1) in patient of FUO | 7th day

SECONDARY OUTCOMES:
Inflammatory marker (TNF) in patient of FUO | 7th day
Inflammatory marker (IL-1) in patient of FUO | 7th day
Inflammatory marker (IL-6) in patient of FUO | 7th day

CONTACTS AND LOCATIONS:
Overall Officials: Chao Wang, Doctor, Study Director — Beijing Friendship Hospital

IPD SHARING:
Plan to Share IPD: No